CLINICAL TRIAL: NCT03198884
Title: A Retrospective Study to Evaluate the Safety and Efficacy of a Nucleoside-Sparing Regimen of Darunavir, Ritonavir, and Dolutegravir
Status: Completed | Type: Observational
Sponsor: Southern Illinois Healthcare Foundation (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, John Verna, Physician Assistant, Southern Illinois Healthcare Foundation
Other Study IDs: 16-1108-100C
Record Dates: First submitted 2017-06-05; First posted 2017-06-26 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Darunavir; Ritonavir; dolutegravir

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Darunavir 800 MG, Norvir 100 MG, Dolutegravir 50 MG

SUMMARY:
A Retrospective Study to Evaluate the Safety and Efficacy of a Nucleoside-Sparing Regimen of Darunavir, Ritonavir, and Dolutegravir

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Received a regimen of darunavir 800 mg/ritonavir 100 mg in combination with dolutegravir 50 mg QD for ≥24 weeks as documented in EMR
* Laboratory reports (CD4, viral load, SrCr) available at time points +/- 4 6 weeks from 12, 24, 36, 48 weeks from start of regimen
* Resistance data (if applicable)

Exclusion Criteria:

* Received a regimen of darunavir/ritonavir in combination with dolutegravir for <24 weeks duration
* Patients receiving darunavir/ritonavir + DTG+NRTI's
* Missing laboratory data in ≥2 study time points
* Patients missing more than five doses over two weeks prior study visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult HIV positive patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-05-01 (Actual)

IPD SHARING:
Plan to Share IPD: No
No plan to share.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A retrospective chart review of appoximately 400 HIV+ patients receiving treatment at an urban diverse FQHC was conducted to identify those who were receiving an NRTI-sparing regimen of DRV and DTG.
Pre-assignment Details: Subjects included were at least 18 years of age, receiving DRV/r + DTG QD for at least 24 weeks and had laboratory data through 48 weeks of follow up. Those excluded were not taking the study regimen, missed more than five doses of medication over two weeks prior to study visit or if there was missing lab data for 2 or more study time points.
Groups:
- Retrospective Chart Review: We conducted a retrospective chart review of approximately 400 HIV+ patients receiving treatment at an urban diverse FQHC to identify those who were receiving a NRTI-sparing regimen of DRV and DTG. Subjects were included if they were ≥ 18 years of age, receiving DRV/r + DTG QD for ≥ 24 weeks, and had laboratory data through 48 weeks of follow up. Subjects were excluded if they received a regimen of DRV/r in combination with DTG for <24 weeks duration, if they received DRV/r + DTG + NRTI's, missed more than five doses over two weeks prior to study visit or if there was missing laboratory data for ≥2 or more study time points. The primary endpoints evaluated were the percent of patients with an RNA <50 copies/mL at 48 weeks after initiation of the regimen, as well as, the change in serum creatinine from baseline to 48 weeks.
Period: Overall Study
Arm/Group | Retrospective Chart Review
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Retrospective Chart Review
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
HIV RNA (copies/mL) [Median (Full Range); unit: copies/mL] — This measurement was conducted at the start and at the conclusion of the study for each participant.
  The range 20 copies/mL to 1,820,101 copies/mL represents the HIV RNA range recorded in study subjects.
  copies/mL | 22.63 [20 to 1,820,101]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With RNA <50 Copies/mL at 48 Weeks
Description: Our first primary endpoint evaluated the percent of study subjects with an RNA <50 copies/mL at 48 weeks after initiation of the once daily two-drug regimen.
Time Frame: 48 weeks
Population: 19 patients meeting the inclusion criteria were analyzed for this study. We evaluated the percentage of study subjects with an HIV RNA < 50 copies at 48 weeks after initiation of the once daily two-drug regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Chart Review
Number analyzed (Participants) | 19
Participants | 19
Statistical Analysis 1: Comparison: Retrospective Chart Review; Test type: Other — The percent of patients with an RNA <50 copies/mL at each time point was analyzed using McNemar's test following the guidelines of the Snapshot algorithm. Missing RNA data was considered a treatment failure. Change in mean serum creatinine from baseline was analyzed using Wilcoxon signed rank test; p < 0.05, McNemar; Change in mean CD4+ cell counts from baseline was analyzed using a paired t-test. All analyses used a p-value of less than or equal to 0.05 as significant. Statistical analyses were performed using R software, version 3.4.3

2. Primary Outcome: The Change in Serum Creatinine From Baseline to 48 Weeks.
Description: A second primary endpoint was evaluating the change in serum creatinine from baseline to 48 weeks for all subjects.
Time Frame: 48 weeks
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Retrospective Chart Review
Number analyzed (Participants) | 20
mg/dL | 73.4 [69.1 to 77.7]
Statistical Analysis 1: Comparison: Retrospective Chart Review; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Mean CD4+ Cell Count From Baseline.
Description: A secondary endpoint included changes from baseline in CD4+ cell counts.
Time Frame: 48 weeks
Population: For week 36 data, 6 study subjects did not have reportable data. These missing data included patient no-shows for labs and lab error (ex, lost sample, insufficient blood/serum drawn to run test).
Measure: Mean (Standard Deviation); unit: cells/μL
Groups:
- Week 24: Data shows mean change in CD4+ cell count (cells/μL) from baseline to week 24.
- Week 36: Data shows mean change in CD4+ cell count (cells/μL) from baseline to week 36.
- Week 48: Data shows mean change in CD4+ cell count (cells/μL) from baseline to week 48.
Arm/Group | Week 24 | Week 36 | Week 48
Number analyzed (Participants) | 20 | 14 | 20
cells/μL | 454 (301) | 428 (254) | 456 (291)

4. Secondary Outcome: Incidence of Adverse Events.
Description: 10 study subjects reported an adverse event.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective Chart Review
Number analyzed (Participants) | 20
Participants
  Insomnia | 6
  Diarrhea | 4
  Headache | 3

5. Secondary Outcome: Number of Grade 1 Adverse Events Reported
Description: 10 study subjects reported adverse events. All adverse events reported (insomnia, diarrhea, headache) were of Grade 1 severity.
  There were no adverse events that led to discontinuation of the study regimen.
Time Frame: 48 weeks
Population: 20 patients were evaluted for adverse events.
Measure: Number; unit: Adverse Events
Groups:
- Adverse Events: As per the studay protocol, an adverse event (AE) is an untoward medical occurence in a patient administered a medicinal product.
Arm/Group | Adverse Events
Number analyzed (Participants) | 20
Adverse Events
  Insomnia | 6
  Diarrhea | 4
  Headache | 3

6. Secondary Outcome: Number of Participants With RNA <50 Copies/mL at 24, 36, and 48 Weeks
Description: This secondary outcome measure analyzed the percentage of subjects with < 50 copies/mL RNA at time points 24, 36 and 48 weeks.
  The percent of subjects with an RNA < 50 copies/mL at each time point was analyzed using McNemar's test following the guidelines of the Snapshot algorithm. Missing RNA data was considered a treatment failure.
Time Frame: 48 weeks
Population: We analyzed data for all participants as indicated in the data table. There was missing data for one study subject at week 24 of the study and missing data for six study subjects at week 36 (blood draws were not completed by patients). Also, data was missing for one study subject at week 48 (blood draw not completed secondary incarceration).
Measure: Count of Participants; unit: Participants
Groups:
- Analysis of HIV RNA at Week 24: At week 24, 75% of subjects had an RNA of < 50 copies/mL. The percent of subjects with an RNA < 50 copies/mL at each time point was analyzed using McNemar's test following the guidelines of the Snapshot algorithm. Missing RNA data was considered a treatment failure.
- Analysis of HIV RNA at Week 36: At week 36, 65% of subjects had an RNA of < 50 copies/mL. The percent of subjects with an RNA < 50 copies/mL at each time point was analyzed using McNemar's test following the guidelines of the Snapshot algorithm. Missing RNA data was considered a treatment failure.
- Analysis of HIV RNA at Week 48: At week 48, 95% of subjects had an RNA of < 50 copies/mL. The percent of subjects with an RNA < 50 copies/mL at each time point was analyzed using McNemar's test following the guidelines of the Snapshot algorithm. Missing RNA data was considered a treatment failure.
Arm/Group | Analysis of HIV RNA at Week 24 | Analysis of HIV RNA at Week 36 | Analysis of HIV RNA at Week 48
Number analyzed (Participants) | 19 | 14 | 19
Participants | 19 | 14 | 19

7. Secondary Outcome: Analysis of Creatinine Clearance at Time Points 24, 36 and 48 Weeks.
Time Frame: 48 weeks
Population: There was missing data for one study subject at week 24 of the study and missing data for six study subjects at week 36 (blood draws were not completed by patients). In addition, data was missing for one study subject at week 48 (blood draw not completed secondary incarceration).
Measure: Mean (Full Range); unit: mg/dL
Groups:
- Analysis of Serum Creatinine at Week 24: There were no significant differences in creatinine clearance from baseline to 24 weeks.
- Analysis of Serum Creatinine at Week 36: There were no significant differences in creatinine clearance from baseline to 36 weeks.
- Analyis of Serum Creatinine at Week 48: There were no significant differences in creatinine clearance from baseline to 48 weeks.
Arm/Group | Analysis of Serum Creatinine at Week 24 | Analysis of Serum Creatinine at Week 36 | Analyis of Serum Creatinine at Week 48
Number analyzed (Participants) | 19 | 14 | 19
mg/dL | 75.8 [56.4 to 95.4] | 69.1 [47.4 to 90.7] | 77.7 [57.0 to 98.5]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for a total of 3 months.
Arm/Group | Retrospective Chart Review
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 10/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retrospective Chart Review (N=20)
insomnia (Nervous system disorders) | 6 (6) — Insomnia
Diarrhea (Gastrointestinal disorders) | 4 (4) — Diarrhea
Headache (Nervous system disorders) | 3 (3) — Headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT03198884/Prot_SAP_000.pdf